CLINICAL TRIAL: NCT07116161
Title: Pilot Study of Exercise Therapy and Cognitive Behavioural Therapy for Fatigue in Female Cancer Patients in Singapore
Brief Title: Exercise Therapy and Cognitive Behavioural Therapy for Fatigue in Female Cancer Patients in Singapore
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore Cancer Society (Other); Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-0016
Record Dates: First submitted 2025-07-07; First posted 2025-08-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Fatigue; Breast Cancer Female
Keywords: Exercise Therapy; Cognitive Behavioural Therapy
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Exercise Therapy Arm (GET) (Experimental)
  Interventions: Other: Graded Exercise Therapy Arm (GET)
- Exercise Therapy (GET) plus Cognitive Behavioural Therapy (CBT) (Experimental)
  Interventions: Other: Experimental: Exercise Therapy (GET) plus Cognitive Behavioural Therapy (CBT)

INTERVENTIONS:
Other: Graded Exercise Therapy Arm (GET) — Consists of a self-supervised individualized exercise prescription by the rehabilitation professional consisting of aerobic (e.g. brisk walking / cycling) and resistance training exercises, customized by patient preference.
  Arms: Graded Exercise Therapy Arm (GET)
Other: Experimental: Exercise Therapy (GET) plus Cognitive Behavioural Therapy (CBT) — Consists of four major components adapted from previous studies,13,15,16 and delivered by qualified and trained study psychologists. First, the ABCD model of cognitive behavioural therapy (A: activating events, B: beliefs, C: consequences, D: Dispute) will be taught and applied to identify negative, unhelpful beliefs and the emotional, behavioural and physical consequences of those beliefs. Second, patients were taught behavioural strategies to manage fatigue (e.g. sleep hygiene, activity scheduling). Lastly, participants will be guided to reformulate dysfunctional cognitions regarding fatigue, improve coping strategies in relation to significant others (e.g. family, friends) and set goals.
  Arms: Exercise Therapy (GET) plus Cognitive Behavioural Therapy (CBT)

SUMMARY:
The purpose of this research study is to investigate the acceptability, feasibility, and effectiveness of exercise therapy and cognitive behavioral therapy (CBT) in improving fatigue levels and breast cancer treatment adherence in breast cancer patients.

DETAILED DESCRIPTION:
This is a randomized controlled, pilot intervention study enrolling 100 female breast cancer patients recruited from National Cancer Centre Singapore, Singapore General Hospital, NCCS Satellite Clinic @ Sengkang General Hospital, and NCCS Satellite Clinic @ Changi General Hospital.

Participants who are deemed eligible by their attending healthcare professional or indicate fatigue on the distress thermometer scale will be referred to the study research assistants or study investigators for further screening. Study research assistants or study investigators will use the Citrix SCM and OAS platform to review patient medical records and appointments.

The study research assistants or study investigators will screen participants based on the study's inclusion and exclusion criteria. They will then approach eligible participants during their clinic appointments or via telephone to introduce the study to them. Interested participants will be further screened and will be asked, "How would you rate your fatigue on a scale of 0 to10 with 0 being 'no fatigue' and 10 being the 'worst possible fatigue'?" (One-item fatigue scale score). The study research assistants or study investigators will record the one-item fatigue scale score for the healthcare professional to review.

If the participant is screened to be eligible, the consent process will be done in clinic or at the participant's home by research assistants and/or study investigators. This will take place either on the same day as their clinic appointment or at another mutually agreed upon date and time in a quiet and conducive room as far as possible. During the consent process, patients are given ample opportunity to ask questions. Participants will be given sufficient time to consider their willingness to participate in the study. Participation in the study will be entirely voluntary. All participants will provide written informed consent prior to their participation in the study.

After obtaining consent, recruited patients will be asked to complete the registration form. They will then be randomized 1:1 into either an exercise therapy arm or an exercise therapy plus CBT arm. They will then complete the baseline questionnaire and the 3 physical function tests, which will be conducted either by a rehabilitation professional, trained research assistant or study investigator. Afterwards, participants will commence the 12-week intervention they have been randomized into (exercise therapy or exercise therapy and CBT). Exercise therapy and CBT will each consist of up to four 1-hour telemedicine sessions using Zoom over 12 weeks, focusing on physical activity and psychosocial elements. The exercise therapy and CBT telemedicine sessions will be arranged at a mutually agreed upon date and time. Follow up visits will be conducted face-to-face in person at the study's site clinics or at the participant's home at a mutually agreed upon date and time at 3 months (Time 1), 6 months (Time 2) and 12 months post-enrolment (Time 3).

At each follow-up visit, the 3 physical function tests [i.e., 6-minute walk test (6MWT), Handgrip strength (HGS), and 5 times sit-to-stand test (5xSTS)] and corresponding follow-up questionnaire (Month 3, Month 6 and Month 12) will be administered by either a rehabilitation professional, trained research assistant or study investigator. The 6-Minute Walk Test (6MWT) is a submaximal exercise test that assesses walking endurance and aerobic capacity. Participants will walk a set circuit for six minutes, and the score is the total distance walked (in metres). The Hand Grip Strength (HGS) test measures isometric strength of the hand and forearm. Participants will sit comfortably with their forearm in a neutral position and elbow at a 90-degree angle, then squeeze a dynamometer as hard as possible with each hand. The average and maximum value (in kilograms) from three trials for each hand will be recorded. The Five Times Sit to Stand (5xSTS) test assesses lower limb strength. Participants will stand up and sit down five times as quickly as possible, and the score is the time (in seconds) to complete the repetitions. Participants are allowed to choose the language of the questionnaires, exercise therapy and CBT sessions (English or Mandarin), which will apply to all questionnaires and sessions. All questionnaires will be administered electronically using FormSG.

Exercise therapy will consist of a self-supervised individualized exercise prescription by the rehabilitation professional consisting of aerobic (e.g. brisk walking / cycling) and resistance training exercises, customized by patient preference. Note that exercise therapy is part of routine clinical care. However, conducting exercise therapy via teleconsulting, while occasionally done based on patient needs, is not considered part of routine clinical care. In the first session, an initial assessment and exercise prescription will be conducted, which will involve evaluating patient's fatigue, reviewing their medical history, setting personalized exercise goals, prescription of low-intensity exercise plan, education on monitoring fatigue and modifying exercises, and a review of the exercise booklet. The first review will take place in the second session, which will involve reviewing the exercise booklet, exercise adherence and fatigue levels, assessing progress in endurance and strength and adjustment of exercises accordingly. Any barriers to exercise and monitoring for new symptoms will also be discussed and addressed. The third and fourth session will be the same as in the second session. However, the fourth session will also cover long-term exercise recommendations and planning for continued independent exercise. The study's research assistants or study investigators will conduct weekly calls to check on adherence to exercises, compliance, and any difficulties or symptoms experienced. The information collected will be entered into a FormSG survey and accessed by rehabilitation professionals, who will provide feedback to the patient via email and/or call. Rehabilitation professional will do four follow-up reviews at each time point (week 0, 4, 8, and 12) during the 12-week intervention period to review the exercises and modify if required. The CBT intervention will have four major components adapted from previous studies and delivered by trained clinical psychologists or psychology trainees under supervision of a clinical psychologist. First, the model of CBT will be taught and applied to identify negative, unhelpful beliefs and the emotional, behavioural and physical consequences of those beliefs. Second, patients were taught behavioural strategies to manage fatigue (e g. sleep hygiene, activity scheduling). Lastly, participants will be guided to reformulate dysfunctional cognitions regarding fatigue, improve coping strategies in relation to significant others (e.g. family, friends) and set goals.

ELIGIBILITY:
Inclusion Criteria:

Primary cohort (N=90):

1. Female
2. ≥21 years of age
3. Stage I-III breast cancer regardless of hormone receptor status or human epidermal growth factor receptor 2 (HER2) status
4. Completed surgery
5. Completed adjuvant chemotherapy, if indicated
6. Reported fatigue (One-item fatigue scale score ≥ 4)
7. Ability to read and communicate in English or Mandarin
8. Willing to provide informed consent for the study participation

Exploratory cohort (N=10):

1. Female
2. ≥21 years of age
3. Stage IV breast cancer regardless of hormone receptor status or human epidermal growth factor receptor 2 (HER2) status
4. Completed surgery
5. Currently receiving systemic therapy (e.g. endocrine therapy, chemotherapy, targeted therapy or immunotherapy)
6. Reported fatigue (One-item fatigue scale score ≥ 4)
7. Ability to read and communicate in English or Mandarin
8. Willing to provide informed consent for the study participation

Exclusion Criteria for both cohorts:

1. Pregnant or lactating
2. Presence of dementia or major psychiatric disease
3. Deemed medically unsuitable by medical team for low to moderate intensity exercise
4. Unable or unwilling for tele-counselling sessions
5. Uncontrolled pain or undiagnosed pain
6. Low blood counts: Hb <8.0, Platelet <50K, ANC <1
7. Electrolyte imbalances: K <3.0, Na <130
8. Cardiovascular diseases, including but not limited to: LVEF <35%, uncontrolled arrhythmias, severe coronary artery disease, severe valvular heart disease, uncontrolled hypertension etc. not cleared by a cardiologist
9. Active infection
10. Currently engaged in moderate to vigorous physical activity

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction with Exercise Therapy and Cognitive Behavioural Therapy (CBT) | Up to 12 months post-enrolment.
  Measured using a 8-item Client Satisfaction Questionnaire. Each item is rated on a 4-point scale, with higher scores indicating greater satisfaction.
Perceived Cultural Sensitivity of the Intervention | Up to 12 months post-enrolment.
  Measured using 4 items adapted from the Cultural Sensitivity Assessment Tool. Each item is rated on a 4 point-scale (1 = Strongly Disagree, 4 = Strongly Agree) with higher scores indicating greater cultural sensitivity.
Uptake and Adherence to Exercise Therapy and Cognitive Behavioural Therapy (CBT) | 3 Months post-enrolment.
  Measured using the percentage of randomized patients who attended at least one session of their allocated intervention and the percentage of randomized patients who completed their allocated interventions.
Willingness to Pay for Therapy Sessions | 3 Months post-enrolment.
  * Measured using a 10-item custom survey based on a step-wise price-point method ($130, $100, $75, $50, $30 per session) to reflect a range of rates covering private and subsidized rates of different tiers.
  * Participants respond with binary Yes/No options, followed by questions assessing willingness to participate if costs are covered by Medisave.
  * This allows estimation of maximum willingness to pay under both cash and insurance-covered scenarios.

SECONDARY OUTCOMES:
Preliminary Effectiveness (Fatigue) | Up to 12 months post-enrolment.
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) subscale evaluates changes in self-reported fatigue levels, a key symptom among breast cancer survivors. FACIT-F scores range from 0 to 52, with higher scores indicating less fatigue.
Adherence to Breast Cancer Treatments | Up to 12 months post-enrolment.
  5-item medication adherence survey adapted from prior studies measuring adherence to prescribed medications over the past 3 months. The primary measure item asks how often participants took their medication as prescribed over the past 3 months. Nonadherence is defined as 75% of the time or less. Additional items assess frequency of forgetting or intentionally skipping medications, with nonadherence defined as once per week or more. Two items address medication switching and discontinuation. Participants who skipped medications only due to switching between tamoxifen and aromatase inhibitors (AIs) will be considered adherent, while those who discontinued tamoxifen or an AI will be asked to provide reasons.
Quality of Life (QoL) | Up to 12 months post-enrolment.
  Functional Assessment of Cancer Therapy - General (FACT-G), assesses quality of life. FACT-G scores range from 0-108 with higher scores indicating better quality of life.
Godin-Shephard Leisure-Time Physical Activity Questionnaire (GLTPAQ) | Up to 12 months post-enrolment.
  Captures the frequency and intensity of participants' physical activity during their free time. GLTPAQ scores are calculated based on frequency and intensity of weekly leisure activity. A score of 24 or more indicates active, a score of 23 or less indicates insufficient activity.
6-Minute Walk Test (6MWT) | Up to 12 months post-enrolment.
  Measures the distance (in metres) an individual can walk in six minutes as an indicator of walking endurance and aerobic capacity
Handgrip Strength (HGS) | Up to 12 months post-enrolment.
  The average and maximum value (in kilograms) from three trials for each hand. Measures the isometric strength of the hand and forearm
5 Times Sit-to-Stand Test (5xSTS) | Up to 12 months post-enrolment.
  Measures the time (in seconds) it takes for a person to rise from a seated position to standing five times in succession, reflecting lower limb strength.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ryan Shea YC TAN, MBBS, MRCP(UK), MMed, Principal Investigator — National Cancer Centre, Singapore
Locations (4):
- Singapore (4):
  - National Cancer Centre, Singapore (NCCS), Singapore
  - Singapore General Hospital, Singapore
  - NCCS Satellite Clinic @ Changi General Hospital, Singapore
  - NCCS Satellite Clinic @ Sengkang General Hospital, Singapore